CLINICAL TRIAL: NCT05283083
Title: Decatecholaminisation With Dexmedetomidine for Reduction of Mortality in Septic Shock: A Randomized Clinical Trial
Brief Title: Decatecholaminisation of Septic Shock With Dexmedetomidine and In-hospital Mortality
Acronym: DECATSepsis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.22.02.1889
Record Dates: First submitted 2022-02-28; First posted 2022-03-16 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Septic Shock; Sepsis
Keywords: dexmedetomidine; randomized controlled trial
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: An open label randomized controlled trial
Masking Description: There is no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine (Experimental): Patients will receive dexmedetomidine infusion according to the protocol plus the usual care.
  We will evaluate patients for inclusion in the study after 6 hours on NE infusion, given stabilization of the MAP > 65 mmHg. In the DEX group, we will commence DEX infusion at the rate of 0.2 mcg.kg-1.h-1 without a loading dose, then titrate DEX infusion to maintain the HR from 60 to 90 bpm.
  Titration of the DEX infusion rate will not be more than 0.1 mcg.kg-1.h-1 every 30 minutes at any time. The maximum DEX infusion rate will be 0.7 mcg.kg-1.h-1.
  We aim to continue DEX infusion for 48 hours. After 48 hours of DEX infusion, we will taper the DEX infusion over one hour.
  According to our protocol, DEX infusion would trigger either STOP events or hemodynamic assessment events:
  Interventions: Drug: Dexmedetomidine
- Usual care without dexmedetomidine infusion (No Intervention): The patients in this group will receive the usual care.

INTERVENTIONS:
Drug: Dexmedetomidine — A highly-selective alpha-2 agonist with sedative, analgesic, and sympatholytic effects.
  Other Names: Precedex, Dexdor, Dexdomitor, Sileo
  Arms: Dexmedetomidine

SUMMARY:
The study aims to determine whether the infusion of DEX in septic shock can reduce in-hospital mortality, norepinephrine infusion, need and duration for mechanical ventilation, and acute kidney injury without significant adverse events.

DETAILED DESCRIPTION:
During septic shock, acute stress response includes neural and humoral autonomic flaring, which tend to be beneficial in the short term. Once shock occurs, it is a failure of the compensation trial. In addition, chronic autonomic stimulation risks myocardial injury, immunosuppression, insulin resistance, and thrombo-embolic tendency.

The investigators hypothesized that dacatecholaminisation with dexmedetomidine - as calibrated by heart rate control - would reduce the in-hospital mortality in septic shock, whether the patient is mechanically ventilated or not. The study aims to determine whether the infusion of DEX in septic shock can reduce in-hospital mortality, norepinephrine infusion, need and duration for mechanical ventilation, and acute kidney injury without significant adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) patients of either sex who develop septic shock with heart rate (HR) > 90 beats per minute (bpm).

We choose the definition of septic shock as the start of norepinephrine (NE) infusion to maintain the mean arterial blood pressure (MAP) of ≥ 65 mmHg in a case of sepsis (≥ 2 SIRS criteria plus suspicion or confirmation of infection).

Exclusion Criteria:

* Patient refusal or inability to obtain consent
* Failure of hemodynamic stabilization or hemoglobin < 7 gm/dl at time of inclusion
* Severe cardiac dysfunction (Ejection Fraction (EF) < 30%)
* History of heart block or patient on pacemaker
* Chronic liver Disease (Child-Pugh classification C)
* Severe valvular heart disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | Through study completion, an average of 3 months
  The investigators will review the patient status on discharge from the hospital, alive or dead

SECONDARY OUTCOMES:
Norepinephrine equivalent dose (NED) | over the first 3 days after enrolment or death, which comes first
  reported as the average of the serial measurements; the NED of epinephrine will be estimated as 1:1 ratio, reported as mcg/kg/min (Shruti Goradia et al, 2021)
Need for epinephrine infusion | over the first 3 days after enrolment or death, which comes first
  Categorical variable (as yes/no outcome)
Heart rate (HR) beat per minute | over the first 3 days after enrolment or death, which comes first
  reported as the average of the serial measurements
Mean arterial blood pressure (MAP) mmHg | over the first 3 days after enrolment or death, which comes first
  reported as the average of the serial measurements
Initiation of invasive mechanical ventilation (IMV) in non-ventilated patients | Through study completion, an average of 3 months
  Categorical variable (as yes/no outcome)
Early acute kidney injury | 48 hours after ICU admission in previously normal kidney function
  Categorical variable (as yes/no outcome) - as defined by Khwaja, A., 2012. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clinical Practice, 120(4), pp.c179-c184.
Late acute kidney injury | 7 days after ICU admission in previously normal kidney function
  Categorical variable (as yes/no outcome) - as defined by the Khwaja, A., 2012. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clinical Practice, 120(4), pp.c179-c184.

CONTACTS AND LOCATIONS:
Overall Officials: Moataz M Emara, MD, EDAIC, Study Director — Mansoura University Faculty of Medicine
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The anonymously patient data will be available on reasonable request - according to the local IRB approval - from the corresponding author and the central study contact, Moataz Emara at mm.emara@mans.edu.eg or mm.emara@yahoo.com.
Time Frame: will be shared shortly.
Access Criteria: The anonymously patient data will be available on reasonable request - according to the local IRB approval - from the corresponding author and the central study contact, Moataz Emara at mm.emara@mans.edu.eg or mm.emara@yahoo.com.

REFERENCES:
- [Derived] Ezz Al-Regal AR, Ramzy EA, Atia AAA, Emara MM. Dexmedetomidine for Reducing Mortality in Patients With Septic Shock: A Randomized Controlled Trial (DecatSepsis). Chest. 2024 Dec;166(6):1394-1405. doi: 10.1016/j.chest.2024.06.3794. Epub 2024 Jul 14. PMID 39004217